CLINICAL TRIAL: NCT04034589
Title: Phase II Study of Pyrotinib in Combination With Fulvestrant in Patients With Human Epidermal Growth Factor Receptor 2 (HER2) Positive，Hormone Receptor（HR）-Positive Metastatic Breast Cancer
Brief Title: Pyrotinib in Combination With Fulvestrant in Patients With HER2 Positive，HR-Positive Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Ying Wang, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-KY-049
Record Dates: First submitted 2019-07-21; First posted 2019-07-26 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pyrotinib plus fulvestrant (Experimental): Pyrotinib(400 mg once daily) + fulvestrant (500 mg, administered on days 0, 14 (plus or minus 3 days), 28 (plus or minus 3 days), and every 28 (plus or minus 3 days) days)
  Interventions: Drug: Pyrotinib combined with fulvestrant

INTERVENTIONS:
Drug: Pyrotinib combined with fulvestrant — Pyrotinib 400 mg once daily; Fulvestrant 500 mg administered on days 0, 14 (plus or minus 3 days), 28 (plus or minus 3 days), and every 28 (plus or minus 3 days) days

SUMMARY:
HR+/HER2+（Human epidermal growth factor receptor 2 positive and hormone receptor positive）metastatic breast cancer is a special subtype of HER2+breast cancer. Conventional guidelines recommend chemotherapy combined with trastuzumab targeted therapy for this subtype of patients. However, the choice of treatment for these patients after treatment progress is a research hotspot in this field. Pyrotinib is a new class I small molecule Tyrosine kinase inhibitors（TKI） drug with high efficacy and low toxicity after the progress of trastuzumab therapy. Fulvestrant is the most preferred single-drug therapy for HR + metastatic breast cancer recommended unanimously by the guidelines, and fulvestrant and small molecule TKI have synergistic effects. Therefore, we envisage that fulvestrant combined with Pyrotinib in the treatment of HR+/HER2+ metastatic breast cancer in clinical practice has the advantages of improving efficacy and survival. To this end, we intend to conduct a prospective, multi-center, phase II clinical trial to evaluate the efficacy and safety of erlotinib in combination with fulvestrant in patients with human epidermal growth factor receptor 2 (HER2) positive，hormone receptor-positive metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed HER2 positive, hormone receptor-positive patients with locally advanced or metastatic breast cancer: HER2 IHC 3+, or HER2 IHC 2+ and FISH detection gene amplification, ER（estrogen receptor） and/or PR（progesterone receptor） Immunohistochemical staining of more than 10% tumor cells)
2. Aged ≥18 and ≤70 years.
3. ECOG（Eastern Cooperative Oncology Group） performance status of 0 to 1.
4. The life expectancy of more than 12 weeks;
5. At least one measurable lesion exists(RECIST 1.1，Response Evaluation Criteria in Solid Tumors ), or only bone metastasis.
6. Previous neoadjuvant or adjuvant use of trastuzumab, but the disease-free interval between the end of the last trastuzumab and the progression of tumors was more than 12 months
7. Trastuzumab has not been treated in the past or only received first-line treatment for metastatic diseases.
8. It is required that previous (neo) adjuvant or endocrine therapy be given to patients, and that progress of the disease occur during or after treatment.
9. Patients with adequate organ function before enrollment:

Neutrophil granulocyte≥1.5×10^9/L Platelet≥100×10^9/L Hemoglobin≥90 g/L Signed informed consent.

Exclusion Criteria:

1. Patients who have not received trastuzumab, chemotherapy or endocrine therapy before;
2. Patients with visceral crisis;
3. Patients unable to swallow, with chronic diarrhea, intestinal obstruction, or multiple factors that affect drug use and absorption;
4. Patients with malignant serous effusion which cannot be controlled by drainage or other methods;
5. Less than 4 weeks from the last treatment in the last clinical trial;
6. Receiving any other antitumor therapy;
7. History of other malignancy within the last 5 years, except for carcinoma in situ of the cervix, basal cell carcinoma or squamous cell carcinoma of the skin that has been previously treated with curative intent;
8. Patients with serious heart disease;
9. Allergy to Pyrotinib; the history of immunodeficiency；
10. Known history of neurological or psychiatric disease, including epilepsy or dementia;
11. Patients during pregnancy or lactation, patients with childbearing potential tested positive in a baseline pregnancy test, or patients unwilling to take effective contraceptive measures throughout the trial;
12. Evidence of significant medical illness that will substantially increase the risk of the participation or completion of the study in the investigator's judgment. Examples included, but not limited to, hypertension, severe diabetes, etc;
13. Patients not eligible for this study judged by the investigator.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2019-07-17 (Actual); Primary Completion 2021-07-06 (Estimated); Study Completion 2022-07-06 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Estimated 12 months
  From enrollment to progression or death (for any reason)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Estimated 12 months
  Ratio of CR and PR in all subjects
Clinical Benefit rate (CBR) | Estimated 12 months
  Ratio of CR,PR and SD greater than or equal to 24 weeks in all subjects
Overall Survival (OS) | Estimated 24 months
  From enrollment to death (for any reason)
Adverse Events and Serious Adverse Events | From informed consent through 28 days following treatment completion
  Safety
Efficacy correlation biomarkers | Estimated 12 months
  Next Generation Gene Sequencing（NGS） detection of tissue specimens to obtain information on drug sensitivity-related biomarkers , eg, PIK3CA, PTEN, TMB，ESR1，ESR2
the quality of life | Estimated 24 months
  All patients need to fill in the Functional Assessment of Cancer Therapy-Breast (FACT-B), a 44-item self-report instrument designed to measure multidimensional quality of life (QL) in patients with breast cancer.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Sun Yat-Sen University Cancer Center, Guangyuan
  - Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou

IPD SHARING:
Plan to Share IPD: No
Individual participant data can be obtained by writing to researchers.

REFERENCES:
- [Background] Xia W, Bacus S, Hegde P, Husain I, Strum J, Liu L, Paulazzo G, Lyass L, Trusk P, Hill J, Harris J, Spector NL. A model of acquired autoresistance to a potent ErbB2 tyrosine kinase inhibitor and a therapeutic strategy to prevent its onset in breast cancer. Proc Natl Acad Sci U S A. 2006 May 16;103(20):7795-800. doi: 10.1073/pnas.0602468103. Epub 2006 May 8. PMID 16682622
- [Background] Kaufman B, Mackey JR, Clemens MR, Bapsy PP, Vaid A, Wardley A, Tjulandin S, Jahn M, Lehle M, Feyereislova A, Revil C, Jones A. Trastuzumab plus anastrozole versus anastrozole alone for the treatment of postmenopausal women with human epidermal growth factor receptor 2-positive, hormone receptor-positive metastatic breast cancer: results from the randomized phase III TAnDEM study. J Clin Oncol. 2009 Nov 20;27(33):5529-37. doi: 10.1200/JCO.2008.20.6847. Epub 2009 Sep 28. PMID 19786670
- [Background] Johnston S, Pippen J Jr, Pivot X, Lichinitser M, Sadeghi S, Dieras V, Gomez HL, Romieu G, Manikhas A, Kennedy MJ, Press MF, Maltzman J, Florance A, O'Rourke L, Oliva C, Stein S, Pegram M. Lapatinib combined with letrozole versus letrozole and placebo as first-line therapy for postmenopausal hormone receptor-positive metastatic breast cancer. J Clin Oncol. 2009 Nov 20;27(33):5538-46. doi: 10.1200/JCO.2009.23.3734. Epub 2009 Sep 28. PMID 19786658
- [Background] Johnston SRD, Hegg R, Im SA, Park IH, Burdaeva O, Kurteva G, Press MF, Tjulandin S, Iwata H, Simon SD, Kenny S, Sarp S, Izquierdo MA, Williams LS, Gradishar WJ. Phase III, Randomized Study of Dual Human Epidermal Growth Factor Receptor 2 (HER2) Blockade With Lapatinib Plus Trastuzumab in Combination With an Aromatase Inhibitor in Postmenopausal Women With HER2-Positive, Hormone Receptor-Positive Metastatic Breast Cancer: ALTERNATIVE. J Clin Oncol. 2018 Mar 10;36(8):741-748. doi: 10.1200/JCO.2017.74.7824. Epub 2017 Dec 15. PMID 29244528 (Retraction: PMID 32822279 J Clin Oncol. 2021 Jan 1;39(1):95)
- [Background] Robertson JFR, Bondarenko IM, Trishkina E, Dvorkin M, Panasci L, Manikhas A, Shparyk Y, Cardona-Huerta S, Cheung KL, Philco-Salas MJ, Ruiz-Borrego M, Shao Z, Noguchi S, Rowbottom J, Stuart M, Grinsted LM, Fazal M, Ellis MJ. Fulvestrant 500 mg versus anastrozole 1 mg for hormone receptor-positive advanced breast cancer (FALCON): an international, randomised, double-blind, phase 3 trial. Lancet. 2016 Dec 17;388(10063):2997-3005. doi: 10.1016/S0140-6736(16)32389-3. Epub 2016 Nov 29. PMID 27908454
- [Background] Robertson JFR, Steger GG, Neven P, Barni S, Gieseking F, Nole F, Pritchard KI, O'Malley FP, Simon SD, Kaufman B, Petruzelka L. Activity of fulvestrant in HER2-overexpressing advanced breast cancer. Ann Oncol. 2010 Jun;21(6):1246-1253. doi: 10.1093/annonc/mdp447. Epub 2009 Oct 29. PMID 19875750
- [Result] Wang YC, Morrison G, Gillihan R, Guo J, Ward RM, Fu X, Botero MF, Healy NA, Hilsenbeck SG, Phillips GL, Chamness GC, Rimawi MF, Osborne CK, Schiff R. Different mechanisms for resistance to trastuzumab versus lapatinib in HER2-positive breast cancers--role of estrogen receptor and HER2 reactivation. Breast Cancer Res. 2011;13(6):R121. doi: 10.1186/bcr3067. Epub 2011 Nov 28. PMID 22123186